CLINICAL TRIAL: NCT04985383
Title: An Open Label Phase 1 Study to Compare the Safety and Tolerability of the AKST1210 Column at Different Blood-Flow Rates in Patients With End-Stage Renal Disease (ESRD) Undergoing Hemodialysis (HD)
Brief Title: Study to Compare Safety and Tolerability of AKST1210 Column at 2 Blood Flow Rates in Subjects With ESRD on Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alkahest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKST1210-101
Record Dates: First submitted 2021-07-01; First posted 2021-08-02 (Actual); Results first posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- AKST1210 device (Experimental): AKST1210 column will be connected in series for the duration of each hemodialysis session.
  Interventions: Device: AKST1210 S-15 at 250 mL/min; Device: AKST1210 S-15 at 450 mL/min; Device: AKST1210 S-25 at 250 mL/min; Device: AKST1210 S-25 at 450 mL/min; Device: AKST1210 S-35 at 250 mL/min; Device: AKST1210 S-35 at 450 mL/min

INTERVENTIONS:
Device: AKST1210 S-15 at 250 mL/min — Procedure: Hemodialysis, AKST1210 column size 150mL and blood-flow rate at 250mL/min
  Other Names: S-15 at 250 mL/min
Device: AKST1210 S-15 at 450 mL/min — Procedure: Hemodialysis, AKST1210 column size 150mL and blood-flow rate at 450mL/min
  Other Names: S-15 up to 450 mL/min
Device: AKST1210 S-25 at 250 mL/min — Procedure: Hemodialysis, AKST1210 column size 250mL and blood-flow rate at 250mL/min
  Other Names: S-25 at 250 mL/min
Device: AKST1210 S-25 at 450 mL/min — Procedure: Hemodialysis, AKST1210 column size 250mL and blood-flow rate at 450mL/min
  Other Names: S-25 at 450 mL/min
Device: AKST1210 S-35 at 250 mL/min — Procedure: Hemodialysis, AKST1210 column size 350mL and blood-flow rate at 250mL/min
  Other Names: S-35 at 250 mL/min
Device: AKST1210 S-35 at 450 mL/min — Procedure: Hemodialysis, AKST1210 column size 350mL and blood-flow rate at 450mL/min
  Other Names: S-35 at 450 mL/min

SUMMARY:
This study is to evaluate the safety and tolerability of the AKST1210 column at blood-flow rates greater than 250 mL/min in subjects with end-stage renal disease (ESRD) undergoing hemodialysis (HD). The study will assess the safety, tolerability, and impact on HD parameters when the AKST1210 column is used at a blood-flow of up to 450 mL/min.

DETAILED DESCRIPTION:
This is an open-label study in approximately 12 to 15 subjects between 40 and 75 years of age with ESRD on HD. The objective of this study is to explore the safety and tolerability of the AKST1210 column at blood-flow rates greater than 250 mL/min in subjects with ESRD undergoing HD. The proposed study will assess the safety, tolerability, and impact on HD parameters when the AKST1210 column is used at a blood-flow rates of up to 450 mL/min. Each participant, per the protocol, will be sequentially treated to each column and blood-flow rate combination.

The incidence of IDH events will be one factor used to determine column size/blood-flow rate escalation/de-escalation as well as discontinuation from the study. The planned duration of subject participation is approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 40 - 75 years, inclusive.
2. End Stage Renal Disease (ESRD) requiring HD.
3. Dialysis vintage ≥ 24 months.
4. Absence of clinically-relevant residual renal function.
5. Regular Hemodialysis (HD) sessions done at blood-flow rates between 400 and 500 mL/min, and with inter-dialysis intervals of 48 hours or more.
6. Stable health status for at least 4 weeks prior to screening based on medical history, and findings from physical examination, laboratory tests, vital signs, and ECG, as assessed by the investigator.
7. Life expectancy > 6 months (as determined by the investigator).
8. Body mass index (BMI) between 18 and 37 kg/m2, inclusive, with a minimum body weight of 52 kg.
9. Must be on stable doses (> 4 weeks) of all treatments for concomitant diseases (e.g., diabetes, hypertension), but this does not apply to medications for conditions related to ESRD (e.g., medications for calcium and phosphate control, anemia).
10. Must be able to follow the study protocol and receive the treatment in the established timeframe.
11. Must provide a signed and dated informed consent form.

Exclusion Criteria:

1. Patients for whom adequate anticoagulation cannot be achieved, such as those with severe anemia, severe hemorrhagic diathesis, severe gastrointestinal ulcers, or who are receiving anticoagulant medications for any reason other than as required for HD. Use of antiplatelet drugs (e.g., aspirin or clopidogrel) is allowed.
2. Patients for whom extracorporeal circulation therapy is contraindicated, such as those with severe cardiac insufficiency, acute myocardial infarction, severe cardiac arrhythmia, acute seizure disorder, or severe uncontrolled hypertension.
3. Patients with Kt/V < 1.2 during recent 8-week period prior to run-in.
4. History of hypersensitivity to heparin, including heparin-induced thrombocytopenia.
5. History of hypersensitivity to the AKST1210 column or its components.
6. Patients who are not anticipated to be able to tolerate blood-flow rates of 450 mL/min during HD (e.g., new vascular access that cannot be used with 14G or 15G needles).
7. Patients who are at higher risk for intradialytic hypotension (IDH) including:

   1. Medical records indicating the occurrence IDH (SBP < 90 mmHg) in more than 30% of HD sessions during a recent 8-week period prior to run-in;
   2. Patients requiring or expected to require extensive fluid management as determined by the investigator;
   3. Presence of pre-dialysis hypotension, defined as SBP < 90 mmHg and/or diastolic blood pressure (DBP) < 50 mmHg, before any of the last 3 dialysis sessions prior to screening;
   4. Diagnosis of IDH in medical records;
   5. Diagnosis of autonomic dysfunction;
   6. Patients who frequently require a ultrafiltration rate (UFR) above 13 mL/kg/h.
8. Patients who are pregnant or breast-feeding or who are planning to become pregnant. Female subjects must not be pregnant or breastfeeding. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and prior to start of treatment. WOCBP and men must agree to use highly-effective contraception (Clinical Trial Facilitation Group 2014) prior to study entry. A woman is considered of childbearing potential following menarche and until becoming postmenopausal (no menses for at least 2 years without an alternative cause). Should a woman become pregnant or suspect she is pregnant while she or her male partner is participating in the study, she should inform her treating physician immediately.
9. Clotting disorders.
10. Sickle cell anemia, hereditary spherocytosis, or autoimmune hemolysis.
11. Clinically significant abnormalities on screening ECG including QT interval corrected for heart rate (QTc) using Fridericia's correction formula [QTcF] of ≥ 500 ms in men and ≥ 520 ms in women.
12. Delirium (encephalopathy).
13. Out of range value for complete blood count (CBC), complete metabolic panel, or coagulation that the investigator deems clinically significant.
14. Thyroid stimulating hormone (TSH) below 0.2 or above 6.0 milli-International unit (mIU)/L, and/or clinically-relevant abnormalities in T3 or T4.
15. Hemoglobin level < 9.0 g/dL.
16. Alanine aminotransferase (ALT) and/or aspartate transaminase (AST) > 3 times upper limit of normal.
17. Uncontrolled type 2 diabetes.
18. Concurrent or have recent participation in another interventional clinical trial. Prior clinical trial subjects must have discontinued investigational agents/devices at least 30 days prior to planned first use of the AKST1210 column.
19. History of severe depression/suicidality requiring hospitalization in the last 6 months.
20. Significant drug or alcohol abuse within the past 12 months.
21. Patients planning to receive renal transplantation during the study.
22. Patients with any other condition and/or situation the investigator believes may interfere with the safety of the subject during study participation, study conduct, or interpretation of study data.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkahest Medical Monitor, Study Director — Alkahest, Inc.
Locations (4):
- United States (4):
  - Renal Consultant Medical Group, Granada Hills, California
  - Valley Renal Medical Group Research, Northridge, California
  - US Renal Care, Gallup, New Mexico
  - US Renal Care - Westover Hills Dialysis, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AKST1210 Device: AKST1210 column will be connected in series for the duration of each hemodialysis session. Participants will progress through 6 weeks of study treatment according to the following device and flow rate combinations:
  Week 1: S-15 at 250 mL/min Week 2: S-15 at up to 450 mL/min Week 3: S-25 at 250 mL/min Week 4: S-25 at up to 450 mL/min Week 5: S-35 at 250 mL/min Week 6: S-35 at up to 450 mL/min
  AKST1210: Procedure: Hemodialysis
Period: Overall Study
Arm/Group | AKST1210 Device
Started | 10
Week 1 AKST1210 S-15 at 250 mL/Min | 9
Week 2 AKST1210 S-15 at up to 450 mL/Min | 9
Week 3 AKST1210 S-25 at 250 mL/Min | 9
Week 4 AKST1210 S-25 at up to 450 mL/Min | 9
Week 5 AKST1210 S-35 at 250 mL/Min | 9
Week 6 AKST1210 S-35 at up to 450 mL/Min | 9
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Safety population includes subjects who received at least 1 (or partial) HD treatment with the AKST1210 column.
Groups:
- AKST1210 Device: AKST1210 column will be connected in series for the duration of each hemodialysis session.
  AKST1210: Procedure: Hemodialysis
Arm/Group | AKST1210 Device
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10
Women of Child Bearing Potential (WOCBP) [Count of Participants; unit: Participants]
  No | 9
  Yes | 1
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.5 (4.07)
Number of Subjects with Baseline Historical IDH Rate [Count of Participants; unit: Participants] — Number of subjects with a baseline historical IDH (intradialytic hypotension/hypotensive) rate (0, 1, 2, 3, and 4) as documented in a subject's medical record during a recent 8-week period prior to the run-in period.
  Participants
    0 | 9
    1 | 1
    2 | 0
    3 | 0
    4 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety as Evaluated by Rate and Severity of Treatment-emergent AEs (TEAEs)
Description: A TEAE is defined as an AE that occurs on or after the date of the first column use.
  Primary and secondary endpoints were assessed at the beginning and end of each week of treatment for a particular column size and blood-flow rate combination (S-15 250 mL/min, S-15 up to 450 mL/min, S-25 250 mL/min, S-25 up to 450 mL/min, S-35 250 mL/min, S-35 up to 450 mL/min). The effect of blood-flow rate was assessed for a given column size as well as intra-subject and across-subject variability.
Time Frame: Screening to Week 7
Population: Safety population: all subjects who received at least 1 (or partial) HD treatment with the AKST1210. NOTE: 10 participants entered the period "AKST1210 S-15 at 250 mL/min," however 9 participants completed all visits in this period and progressed to the following week "AKST1210 S-15 at up to 450 mL/min."
Measure: Count of Participants; unit: Participants
Groups:
- S-15 at 250 mL/Min: AKST1210 column size 150mL and blood-flow rate at 250mL/min
- S-15 at 450 mL/Min: AKST1210 column size 150mL and blood-flow rate at 450mL/min
- S-25 at 250 mL/Min: AKST1210 column size 250mL and blood-flow rate at 250mL/min
- S-25 at 450 mL/Min: AKST1210 column size 250mL and blood-flow rate at 450mL/min
- S-35 at 250 mL/Min: AKST1210 column size 350mL and blood-flow rate at 250mL/min
- S-35 at 450 mL/Min: AKST1210 column size 350mL and blood-flow rate at 450mL/min
Arm/Group | S-15 at 250 mL/Min | S-15 at 450 mL/Min | S-25 at 250 mL/Min | S-25 at 450 mL/Min | S-35 at 250 mL/Min | S-35 at 450 mL/Min
Number analyzed (Participants) | 10 | 9 | 9 | 9 | 9 | 9
Participants
  Severity - Mild | 1 | 0 | 0 | 0 | 0 | 0
  Severity - Moderate | 1 | 0 | 0 | 1 | 0 | 1
  Severity - Severe | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Safety as Evaluated by the Number of Subjects With Intradialytic Hypotensive (IDH) Events
Description: The number and percentage of subjects with Intradialytic Hypotensive (IDH) event(s) summarized by column size and blood-flow rate combination.
  Primary and secondary endpoints were assessed at the beginning and end of each week of treatment for a particular column size and blood-flow rate combination (S-15 250 mL/min, S-15 up to 450 mL/min, S-25 250 mL/min, S-25 up to 450 mL/min, S-35 250 mL/min, S-35 up to 450 mL/min). The effect of blood-flow rate was assessed for a given column size as well as intra-subject and across-subject variability.
Time Frame: Week 1 - S-15 at 250 mL/min, Week 2 - S-15 at up to 450 mL/min, Week 3 - S-25 at 250 mL/min, Week 4 - S-25 at up to 450 mL/min, Week 5 - S-35 at 250 mL/min, Week 6 - S-35 at up to 450 mL/min
Population: Safety population: all subjects who received at least 1 (or partial) HD treatment with the AKST1210 column. NOTE: 10 participants entered the period "AKST1210 S-15 at 250 mL/min," however 9 participants completed all visits in this period and progressed to the following week "AKST1210 S-15 at up to 450 mL/min."
Measure: Count of Participants; unit: Participants
Arm/Group | S-15 at 250 mL/Min | S-15 at 450 mL/Min | S-25 at 250 mL/Min | S-25 at 450 mL/Min | S-35 at 250 mL/Min | S-35 at 450 mL/Min
Number analyzed (Participants) | 10 | 9 | 9 | 9 | 9 | 9
Participants | 1 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Safety as Evaluated by Changes in Total Hemoglobin (Hgb)
Description: Changes in post-HD total hemoglobin at baseline (i.e., the last non-missing value prior to the start of HD with the AKST1210 column) and each scheduled post-baseline timepoint summarized by each column size and blood-flow rate combination.
Time Frame: Baseline, Week 1 - S-15 at 250 mL/min, Week 2 - S-15 at up to 450 mL/min, Week 5 - S-35 at 250 mL/min, Week 6 - S-35 at up to 450 mL/min
Population: Safety population: all subjects who received at least 1 (or partial) HD treatment with the AKST1210 column. Subjects with missing Hgb data ( S-24 at 250mL/min and S-25 at 450mL/min) are excluded from the number analyzed. NOTE: 10 participants entered the period "AKST1210 S-15 at 250 mL/min," however 9 participants completed all visits in this period and progressed to the following week "AKST1210 S-15 at up to 450 mL/min."
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | S-15 at 250 mL/Min | S-15 at 450 mL/Min | S-35 at 250 mL/Min | S-35 at 450 mL/Min
Number analyzed (Participants) | 10 | 9 | 9 | 9
mg/dL | 4.9 (10.76) | 2.2 (9.06) | -4.3 (11.53) | -7.1 (14.86)

4. Primary Outcome: Safety as Evaluated by Changes in Free Hemoglobin (Hgb)
Description: Changes in post-HD free hemoglobin at baseline (i.e., the last non-missing value prior to the start of HD with the AKST1210 column) and each scheduled post-baseline timepoint summarized by each column size and blood-flow rate combination.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | S-15 at 250 mL/Min | S-15 at 450 mL/Min | S-35 at 250 mL/Min | S-35 at 450 mL/Min
Number analyzed (Participants) | 10 | 9 | 9 | 9
mg/dL | 3.4 (8.04) | 1.5 (12.34) | 49.0 (123.87) | 8.7 (15.45)

5. Secondary Outcome: Adequacy of Hemodialysis Measured With Kt/V
Description: Kt/V summarized at baseline and by each column size and flow-rate combination. Kt/V is calculated with Daugirdas' formula from the pre-dialysis to post-dialysis urea nitrogen ratio (R), the weight loss (UF), session length in hours (t), and anthropometric or modeled volume (V) using the equation: Kt/V = In (R - 0.008 x t) + (4 - 3.5 x R) x 0.55 UF/V.
Time Frame: as for outcome 2
Population: Evaluable population: all subjects who completed blood-flow rates up to 450 mL/min for at least 1 column size (e.g., S-15 at 250 and up to 450 mL/min). The number analyzed within each row reflects the available data that was collected for subjects during each treatment period. Subjects with missing Kt/v data are excluded from the number analyzed.
Measure: Mean (Standard Deviation); unit: Kt/V
Groups:
- S-35 at 450 mL/Min: AKST1210 column size 350mL and blood-flow rate at 250mL/min
Arm/Group | S-15 at 250 mL/Min | S-15 at 450 mL/Min | S-25 at 250 mL/Min | S-25 at 450 mL/Min | S-35 at 250 mL/Min | S-35 at 450 mL/Min
Number analyzed (Participants) | 9 | 8 | 7 | 8 | 9 | 8
Kt/V | 1.3 (0.21) | 1.8 (0.28) | 1.2 (0.21) | 1.6 (0.43) | 1.4 (0.25) | 1.6 (0.15)

6. Secondary Outcome: Adequacy of Hemodialysis Measured by Urea Reduction Ratio (URR)
Description: Weekly URR (%) measurements calculated as URR (%) = (1 - post-dialysis BUN / pre-dialysis BUN) * 100 and summarized by each column size and flow-rate combination. Pre-dialysis BUN and Post-Dialysis BUN are hemodialysis values observed within the same dialysis session. URR is a measure of the proportionate reduction in blood urea nitrogen over the course of dialysis.
Time Frame: as for outcome 2
Population: Evaluable population: all subjects who completed blood-flow rates up to 450 mL/min for at least 1 column size (e.g., S-15 at 250 and up to 450 mL/min). The number analyzed within each row reflects the available data that was collected for subjects during each treatment period. Subjects with missing URR data are excluded from the number analyzed.
Measure: Mean (Standard Deviation); unit: URR percentage
Arm/Group | S-15 at 250 mL/Min | S-15 at 450 mL/Min | S-25 at 250 mL/Min | S-25 at 450 mL/Min | S-35 at 250 mL/Min | S-35 at 450 mL/Min
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 6 | 7
URR percentage | 66.2 (3.95) | 77.1 (3.95) | 55.0 (25.00) | 74.1 (11.75) | 68.2 (3.13) | 75.0 (3.05)

7. Secondary Outcome: Total Fluid Balance for Each Column-Size Blood-Flow Rate Combination
Description: Actual fluid removal is calculated as follows: Weight (kg) - Weight Post-Dialysis (kg) and subsequently converting weight to volume (1 kg = 1000 mL).
  Each week contains 3 visits, as indicated in the following parentheses:
  Week 1 - S-15 at 250 mL/min: Visit 5 (Visit #1), Visit 6 (Visit #2), Visit 7 (Visit #3) Week 2 - S-15 at up to 450 mL/min: Visit 8 (Visit #1), Visit 9 (Visit #2), Visit 10 (Visit #3) Week 3 - S-25 at 250 mL/min: Visit 11 (Visit #1), Visit 12 (Visit #2), Visit 13 (Visit #3) Week 4 - S-25 at up to 450 mL/min: Visit 14 (Visit #1), Visit 15 (Visit #2), Visit 16 (Visit #3) Week 5 - S-35 at 250 mL/min: Visit 17 (Visit #1), Visit 18 (Visit #2), Visit 19 (Visit #3) Week 6 - S-35 at up to 450 mL/min: Visit 20 (Visit #1), Visit 21 (Visit #2), Visit 22 (Visit #3)
Time Frame: as for outcome 2
Population: Evaluable population: all subjects who completed blood-flow rates up to 450 mL/min for at least 1 column size (e.g., S-15 at 250 and up to 450 mL/min).
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | S-15 at 250 mL/Min | S-15 at 450 mL/Min | S-25 at 250 mL/Min | S-25 at 450 mL/Min | S-35 at 250 mL/Min | S-35 at 450 mL/Min
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
mL
  Visit #1 | 2144.4 (559.27) | 2288.9 (991.77) | 1933.3 (1065.36) | 2344.4 (1143.58) | 2100.0 (796.87) | 2566.7 (890.22)
  Visit #2 | 1711.1 (1085.64) | 1955.6 (970.97) | 1888.9 (470.22) | 1855.6 (907.07) | 2222.2 (924.36) | 2100.0 (680.07)
  Visit #3 | 2588.9 (814.62) | 2233.3 (1206.23) | 2822.2 (948.39) | 2288.9 (1076.39) | 2500.0 (873.21) | 2355.6 (935.56)

8. Secondary Outcome: Number of Participants Who Achieved the Dry Weight Goal
Description: Number of subjects who were able to achieve the dry weight goal during the allotted HD duration for each visit and column size and blood-flow rate combination.
  Each week contains 3 visits, as indicated in the following parentheses:
  Week 1 - S-15 at 250 mL/min: Visit 5 (Visit #1), Visit 6 (Visit #2), Visit 7 (Visit #3) Week 2 - S-15 at up to 450 mL/min: Visit 8 (Visit #1), Visit 9 (Visit #2), Visit 10 (Visit #3) Week 3 - S-25 at 250 mL/min: Visit 11 (Visit #1), Visit 12 (Visit #2), Visit 13 (Visit #3) Week 4 - S-25 at up to 450 mL/min: Visit 14 (Visit #1), Visit 15 (Visit #2), Visit 16 (Visit #3) Week 5 - S-35 at 250 mL/min: Visit 17 (Visit #1), Visit 18 (Visit #2), Visit 19 (Visit #3) Week 6 - S-35 at up to 450 mL/min: Visit 20 (Visit #1), Visit 21 (Visit #2), Visit 22 (Visit #3)
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | S-15 at 250 mL/Min | S-15 at 450 mL/Min | S-25 at 250 mL/Min | S-25 at 450 mL/Min | S-35 at 250 mL/Min | S-35 at 450 mL/Min
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
Participants
  Visit #1 | 4 | 4 | 2 | 5 | 5 | 4
  Visit #2 | 4 | 5 | 2 | 4 | 6 | 4
  Visit #3 | 4 | 5 | 2 | 3 | 1 | 2

9. Secondary Outcome: Plasma Beta-2 Microglobulin (b2M) Concentrations (Before and After HD) and Contribution of the AKST1210 Column to b2M Removal at Each Column Size and Blood-flow Rate
Description: Least-squares mean arterial ratios (end-HD/pre-HD) and associated 95% confidence intervals (CIs) were determined from a Mixed Model Repeated Measure (MMRM) for the end-HD/pre-HD arterial ratio in the logarithmic scale, with visits (V7, V10, V13, V16, V19, and V22) as a fixed effect, a covariate for baseline b2M protein levels, and a random intercept and covariate for investigational site (or dialyzer type). Note: Visits correspond to blood-flow rate and column combinations.
Time Frame: Week 1 (V7) - S-15 at 250 mL/min, Week 2 (V10) - S-15 at up to 450 mL/min, Week 3 (V13) - S-25 at 250 mL/min, Week 4 (V16) - S-25 at up to 450 mL/min, Week 5 (V19) - S-35 at 250 mL/min, Week 6 (V22) - S-35 at up to 450 mL/min
Population: The b2M Population consists of a subset of the evaluable population that excludes any subjects with Major Protocol Deviations pertaining to blood flow rate as well as any subjects who have documented blood flow rate deviations exceeding +/- 20 mL/min of the protocol-specified blood flow rate at Visits 4, 7, 10, 13, 16, 19 and/or 22.
Measure: Least Squares Mean (95% Confidence Interval); unit: log ratio (mg/L)
Arm/Group | S-15 at 250 mL/Min | S-15 at 450 mL/Min | S-25 at 250 mL/Min | S-25 at 450 mL/Min | S-35 at 250 mL/Min | S-35 at 450 mL/Min
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7
log ratio (mg/L) | -0.9 [-1.2 to -0.6] | -1.0 [-1.3 to -0.7] | -0.8 [-1.1 to -0.5] | -1.1 [-1.4 to -0.9] | -0.9 [-1.2 to -0.6] | -1.3 [-1.6 to -1.0]

10. Secondary Outcome: Number of Occurrences of Visible Thrombosis (Clotting) in the AKST1210 Column, Dialyzer, and/or Tubing
Description: Number of occurrences of visible thrombosis (clotting) in the AKST1210 column, dialyzer, and/or tubing by column size and blood-flow rate combination.
Time Frame: as for outcome 2
Population: Safety population: all subjects who received at least 1 (or partial) HD treatment with the LIXELLE column. NOTE: 10 participants entered the period "AKST1210 S-15 at 250 mL/min," however 9 participants completed all visits in this period and progressed to the following week "AKST1210 S-15 at up to 450 mL/min."
Measure: Count of Participants; unit: Participants
Arm/Group | S-15 at 250 mL/Min | S-15 at 450 mL/Min | S-25 at 250 mL/Min | S-25 at 450 mL/Min | S-35 at 250 mL/Min | S-35 at 450 mL/Min
Number analyzed (Participants) | 10 | 9 | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Plasma Levels of Complement Factors, Including Total Complement CH50, Soluble Complement SC5b-9, and Complement C5a
Description: Plasma levels of complement factors, including total CH50, SC5b-9, and C5a, are summarized by visit for combined column size and blood-flow rate combinations.
Time Frame: Baseline, Week 1 - S-15 at 250 mL/min, Week 6 - S-35 at up to 450 mL/min
Population: Evaluable population: all subjects who completed blood-flow rates up to 450 mL/min for at least 1 column size (e.g., S-15 at 250 and up to 450 mL/min). All column size/blood-flow rate are included in this analysis population.
  NOTE: 10 participants entered the period "AKST1210 S-15 at 250 mL/min," however 9 participants completed all visits in this period and progressed to the following week "AKST1210 S-15 at up to 450 mL/min."
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | AKST1210 Device
Number analyzed (Participants) | 10
g/L
  CH50, Baseline Post-HD | 67.4 (12.14)
  CH50, Visit 7 Post-HD: number analyzed (Participants) | 9
  CH50, Visit 7 Post-HD | 63.6 (13.89)
  CH50, Visit 22 Post-HD: number analyzed (Participants) | 9
  CH50, Visit 22 Post-HD | 61.5 (13.43)
  SC5b-9, Baseline Post-HD: number analyzed (Participants) | 9
  SC5b-9, Baseline Post-HD | 296.7 (101.59)
  SC5b-9, Visit 7 Post-HD: number analyzed (Participants) | 9
  SC5b-9, Visit 7 Post-HD | 624.2 (157.34)
  SC5b-9, Visit 22 Post-HD: number analyzed (Participants) | 9
  SC5b-9, Visit 22 Post-HD | 896.7 (209.87)
  C5a, Baseline Post-HD: number analyzed (Participants) | 9
  C5a, Baseline Post-HD | 9.5 (3.97)
  C5a, Visit 7 Post-HD: number analyzed (Participants) | 9
  C5a, Visit 7 Post-HD | 9.5 (4.08)
  C5a, Visit 22 Post-HD: number analyzed (Participants) | 9
  C5a, Visit 22 Post-HD | 8.9 (1.99)

12. Secondary Outcome: Plasma Levels of Other Proteins, Including Insulin and Adrenocorticotropic Hormone (ACTH)
Description: Plasma levels of other proteins, including insulin and ACTH, at each schedule timepoint summarized by visit for combined column size and blood-flow rate combination.
Time Frame: Baseline, Week 1 - S-15 at 250 mL/min, Week 6 - S-35 at up to 450 mL/min
Population: Evaluable population: all subjects who completed blood-flow rates up to 450 mL/min for at least 1 column size (e.g., S-15 at 250 and up to 450 mL/min). All column size/blood-flow rate are included in this analysis population.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | AKST1210 Device
Number analyzed (Participants) | 10
pmol/L
  Insulin, Baseline Post HD | 87.7 (76.23)
  Insulin, Visit 7 Post HD: number analyzed (Participants) | 9
  Insulin, Visit 7 Post HD | 64.4 (43.80)
  Insulin, Visit 22 Post HD: number analyzed (Participants) | 9
  Insulin, Visit 22 Post HD | 35.2 (13.43)
  ACTH, Baseline Post HD | 11.1 (7.79)
  ACTH, Visit 7 Post HD: number analyzed (Participants) | 9
  ACTH, Visit 7 Post HD | 8.9 (6.19)
  ACTH, Visit 22 Post HD: number analyzed (Participants) | 9
  ACTH, Visit 22 Post HD | 8.7 (10.37)

13. Secondary Outcome: Plasma Levels of Other Proteins, Including Insulin-Like Growth Factor Binding Prot1 (IGFBP1)
Description: Plasma levels of other proteins, including IGFBP1, at each schedule timepoint summarized by visit for combined column size and blood-flow rate combination.
Time Frame: Baseline, Week 1 - S-15 at 250 mL/min, Week 6 - S-35 at up to 450 mL/min
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | AKST1210 Device
Number analyzed (Participants) | 10
ug/L
  IGFBP1, Baseline Post HD | 86.5 (66.62)
  IGFBP1, Visit 7 Post HD: number analyzed (Participants) | 9
  IGFBP1, Visit 7 Post HD | 92.6 (66.19)
  IGFBP1, Visit 22 Post HD: number analyzed (Participants) | 9
  IGFBP1, Visit 22 Post HD | 114.7 (91.38)

ADVERSE EVENTS:
Time Frame: Approximately 12 weeks (up to 4 weeks for screening and 8 weeks on study, inclusive of the 1-week run-in period)
Description: Safety population includes all subjects who received at least 1 (or partial) HD treatment with the LIXELLE column. NOTE: 10 participants entered the period "AKST1210 S-15 at 250 mL/min," however 9 participants completed all visits in this period and progressed to the following week "AKST1210 S-15 at up to 450 mL/min."
Groups:
- Screening/Run-in: No AKST1210 column will be used during the Screening/Run-in period.
  Procedure: Hemodialysis
- AKST1210 S-15 at 250 mL/Min: AKST1210 column size 150mL and blood-flow rate at 250mL/min
- AKST1210 S-15 at up to 450 mL/Min: AKST1210 column size 150mL and blood-flow rate at 450mL/min
- AKST1210 S-25 at 250 mL/Min: AKST1210 column size 250mL and blood-flow rate at 250mL/min
- AKST1210 S-25 at up to 450 mL/Min: AKST1210 column size 250mL and blood-flow rate at 450mL/min
- AKST1210 S-35 at 250 mL/Min: AKST1210 column size 350mL and blood-flow rate at 250mL/min
- AKST1210 S-35 at up to 450 mL/Min: AKST1210 column size 350mL and blood-flow rate at 450mL/min
Arm/Group | Screening/Run-in | AKST1210 S-15 at 250 mL/Min | AKST1210 S-15 at up to 450 mL/Min | AKST1210 S-25 at 250 mL/Min | AKST1210 S-25 at up to 450 mL/Min | AKST1210 S-35 at 250 mL/Min | AKST1210 S-35 at up to 450 mL/Min
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 2/10 | 2/10 | 0/9 | 0/9 | 1/9 | 0/9 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Screening/Run-in (N=10) | AKST1210 S-15 at 250 mL/Min (N=10) | AKST1210 S-15 at up to 450 mL/Min (N=9) | AKST1210 S-25 at 250 mL/Min (N=9) | AKST1210 S-25 at up to 450 mL/Min (N=9) | AKST1210 S-35 at 250 mL/Min (N=9) | AKST1210 S-35 at up to 450 mL/Min (N=9)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dialysis hypotension (Vascular disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
After the study was closed, unreliable data was identified at a single study site and has not been presented here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement contains language that restricts the PI from discussing or publishing Sponsor confidential and/or proprietary information. The embargo period may be extended by mutual agreement of the Sponsor and PI.

DOCUMENTS (2):
  • Study Protocol (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT04985383/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT04985383/SAP_001.pdf